CLINICAL TRIAL: NCT00149162
Title: Multicenter Protocol in Treating Patients With Childhood Acute Myeloid Leukemia. Randomized Study of Maintenance Treatment With Interleukin-2
Brief Title: Treating Patients With Childhood Acute Myeloid Leukemia With Interleukin-2
Acronym: Elam02
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Chiron Corporation (Industry)
Responsible Party: Therese Ngoue, Direction Interregionale de la Recherche Clinique, Ile de France, APHP
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P030441; AOM 03142
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2009-02-12 (Estimated); Status verified 2009-02

CONDITIONS: Leukemia
Keywords: Controlled; Multicenter; International; Randomized study; Direct individual benefit; complete remission after chemotherapy; non allogeneic transplanted
MeSH Terms: conditions — Leukemia | interventions — aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Patients treated by Proleukin
  Interventions: Drug: proleukin
- 2 (No Intervention): Without Proleukin

INTERVENTIONS:
Drug: proleukin — One cycle of treatment : D1 : 2.5 MUI/m2 (subcutaneous); D2 to D5 : 5 MUI / m2 (subcutaneous)
  1 cycle of treatment each month during 12 months
  Other Names: Proleukin = Interleukin II
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the interest of maintenance treatment with interleukin-2 by randomizing the patients being not allogeneic transplanted in complete remission after induction and consolidation chemotherapy concerning the event free survival.

DETAILED DESCRIPTION:
We designed an open randomized study to evaluate the interest of maintenance treatment with interleukin-2 by randomizing the patients being not allogeneic transplanted in complete remission after induction and consolidation chemotherapy concerning the event free survival. A total of 580 patients will be accrued over 7 years. Treatment consists in subcutaneous application of interleukin-2 in treating patients with complete remission by a monthly regimen of 5 days during 1 year after having received a chemotherapy consisting of 1 induction and 3 consolidation treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age: 0 to 18 years
* Prior untreated acute myeloid leukemia (AML) of following cytological types : FAB M0, M1, M2, M4, M4 eosinophil, M5, M6, M7, without FAB classification or showing myelodysplasia (blasts > 20 %)
* Isolated myeloid sarcoma
* Achieved complete remission
* No HLA identical family donor, except for the patients with t(8;21)
* No contraindication for the use of interleukin-2

Exclusion Criteria:

* Trisomy 21
* Promyelocytic leukemia (M3) or M3 variations
* Secondary AML

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 580 (Estimated)
Dates: Start 2005-03; Primary Completion 2010-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Interest of interleukin-2 in complete remission after induction and consolidation chemotherapy concerning the event free survival (event = relapse of toxic death) | 1 year

SECONDARY OUTCOMES:
Analyze the whole toxicity of the regimen | 1 year
Examine the prognostic biological factors | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Guy Leverger, M.D., Principal Investigator — Department of Pediatrics Hematology, Children Armand Trousseau Hospital, 26 Avenue Arnold Netter, 75012 Paris
Locations (1):
- Children Armand Trousseau Hospital, Paris, France

REFERENCES:
- [Background] Lie SO, Jonmundsson G, Mellander L, Siimes MA, Yssing M, Gustafsson G. A population-based study of 272 children with acute myeloid leukaemia treated on two consecutive protocols with different intensity: best outcome in girls, infants, and children with Down's syndrome. Nordic Society of Paediatric Haematology and Oncology (NOPHO). Br J Haematol. 1996 Jul;94(1):82-8. doi: 10.1046/j.1365-2141.1996.d01-1761.x. PMID 8757513
- [Background] Wells RJ, Woods WG, Buckley JD, Odom LF, Benjamin D, Bernstein I, Betcher D, Feig S, Kim T, Ruymann F, et al. Treatment of newly diagnosed children and adolescents with acute myeloid leukemia: a Childrens Cancer Group study. J Clin Oncol. 1994 Nov;12(11):2367-77. doi: 10.1200/JCO.1994.12.11.2367. PMID 7964952
- [Background] Lipshultz SE, Colan SD, Gelber RD, Perez-Atayde AR, Sallan SE, Sanders SP. Late cardiac effects of doxorubicin therapy for acute lymphoblastic leukemia in childhood. N Engl J Med. 1991 Mar 21;324(12):808-15. doi: 10.1056/NEJM199103213241205. PMID 1997853
- [Background] Mertens AC, Wen W, Davies SM, Steinbuch M, Buckley JD, Potter JD, Robison LL. Congenital abnormalities in children with acute leukemia: a report from the Children's Cancer Group. J Pediatr. 1998 Nov;133(5):617-23. doi: 10.1016/s0022-3476(98)70100-3. PMID 9821417
- [Background] Krischer JP, Epstein S, Cuthbertson DD, Goorin AM, Epstein ML, Lipshultz SE. Clinical cardiotoxicity following anthracycline treatment for childhood cancer: the Pediatric Oncology Group experience. J Clin Oncol. 1997 Apr;15(4):1544-52. doi: 10.1200/JCO.1997.15.4.1544. PMID 9193351
- [Background] Behar C, Suciu S, Benoit Y, Robert A, Vilmer E, Boutard P, Bertrand Y, Lutz P, Ferster A, Tokaji E, Manel AM, Solbu G, Otten J. Mitoxantrone-containing regimen for treatment of childhood acute leukemia (AML) and analysis of prognostic factors: results of the EORTC Children Leukemia Cooperative Study 58872. Med Pediatr Oncol. 1996 Mar;26(3):173-9. doi: 10.1002/(SICI)1096-911X(199603)26:33.0.CO;2-H. PMID 8544799
- [Background] Burnett AK, Goldstone AH, Stevens RM, Hann IM, Rees JK, Gray RG, Wheatley K. Randomised comparison of addition of autologous bone-marrow transplantation to intensive chemotherapy for acute myeloid leukaemia in first remission: results of MRC AML 10 trial. UK Medical Research Council Adult and Children's Leukaemia Working Parties. Lancet. 1998 Mar 7;351(9104):700-8. doi: 10.1016/s0140-6736(97)09214-3. PMID 9504514
- [Background] Byrd JC, Dodge RK, Carroll A, Baer MR, Edwards C, Stamberg J, Qumsiyeh M, Moore JO, Mayer RJ, Davey F, Schiffer CA, Bloomfield CD. Patients with t(8;21)(q22;q22) and acute myeloid leukemia have superior failure-free and overall survival when repetitive cycles of high-dose cytarabine are administered. J Clin Oncol. 1999 Dec;17(12):3767-75. doi: 10.1200/JCO.1999.17.12.3767. PMID 10577848
- [Background] Cortes JE, Kantarjian HM, O'Brien S, Giles F, Keating MJ, Freireich EJ, Estey EH. A pilot study of interleukin-2 for adult patients with acute myelogenous leukemia in first complete remission. Cancer. 1999 Apr 1;85(7):1506-13. PMID 10193940
- [Background] Creutzig U, Ritter J, Zimmermann M, Reinhardt D, Hermann J, Berthold F, Henze G, Jurgens H, Kabisch H, Havers W, Reiter A, Kluba U, Niggli F, Gadner H. Improved treatment results in high-risk pediatric acute myeloid leukemia patients after intensification with high-dose cytarabine and mitoxantrone: results of Study Acute Myeloid Leukemia-Berlin-Frankfurt-Munster 93. J Clin Oncol. 2001 May 15;19(10):2705-13. doi: 10.1200/JCO.2001.19.10.2705. PMID 11352963
- [Background] Foa R, Caretto P, Fierro MT, Bonferroni M, Cardona S, Guarini A, Lista P, Pegoraro L, Mandelli F, Forni G, et al. Interleukin 2 does not promote the in vitro and in vivo proliferation and growth of human acute leukaemia cells of myeloid and lymphoid origin. Br J Haematol. 1990 May;75(1):34-40. doi: 10.1111/j.1365-2141.1990.tb02613.x. PMID 2375921
- [Background] Leblanc T, Berger R. Molecular cytogenetics of childhood acute myelogenous leukaemias. Eur J Haematol. 1997 Jul;59(1):1-13. doi: 10.1111/j.1600-0609.1997.tb00953.x. PMID 9260575
- [Background] Maraninchi D, Blaise D, Viens P, Brandely M, Olive D, Lopez M, Sainty D, Marit G, Stoppa AM, Reiffers J, et al. High-dose recombinant interleukin-2 and acute myeloid leukemias in relapse. Blood. 1991 Nov 1;78(9):2182-7. PMID 1932739
- [Background] Meloni G, Foa R, Vignetti M, Guarini A, Fenu S, Tosti S, Tos AG, Mandelli F. Interleukin-2 may induce prolonged remissions in advanced acute myelogenous leukemia. Blood. 1994 Oct 1;84(7):2158-63. PMID 7919330
- [Background] Michel G, Leverger G, Leblanc T, Nelken B, Baruchel A, Landman-Parker J, Thuret I, Bergeron C, Bordigoni P, Esperou-Bourdeau H, Perel Y, Vannier JP, Schaison G. Allogeneic bone marrow transplantation vs aggressive post-remission chemotherapy for children with acute myeloid leukemia in first complete remission. A prospective study from the French Society of Pediatric Hematology and Immunology (SHIP). Bone Marrow Transplant. 1996 Feb;17(2):191-6. PMID 8640165
- [Background] Michel G, Baruchel A, Tabone MD, Nelken B, Leblanc T, Thuret I, Bordigoni P, Bergeron C, Esperou-Bourdeau H, Perel Y, Vannier JP, De Lumley L, Dommergues JP, Lamagnere JP, Couillaud G, Auvrignon A, Schaison G, Leverger G. Induction chemotherapy followed by allogeneic bone marrow transplantation or aggressive consolidation chemotherapy in childhood acute myeloblastic leukemia. A prospective study from the French Society of Pediatric Hematology and Immunology (SHIP). Hematol Cell Ther. 1996 Apr;38(2):169-76. doi: 10.1007/s00282-996-0169-7. PMID 8931998
- [Background] Oshimi K, Oshimi Y, Akutsu M, Takei Y, Saito H, Okada M, Mizoguchi H. Cytotoxicity of interleukin 2-activated lymphocytes for leukemia and lymphoma cells. Blood. 1986 Oct;68(4):938-48. PMID 3489494
- [Background] Perel Y, Auvrignon A, Leblanc T, Vannier JP, Michel G, Nelken B, Gandemer V, Schmitt C, Lamagnere JP, De Lumley L, Bader-Meunier B, Couillaud G, Schaison G, Landman-Parker J, Thuret I, Dalle JH, Baruchel A, Leverger G; Group LAME of the French Society of Pediatric Hematology and Immunology. Impact of addition of maintenance therapy to intensive induction and consolidation chemotherapy for childhood acute myeloblastic leukemia: results of a prospective randomized trial, LAME 89/91. Leucamie Aique Myeloide Enfant. J Clin Oncol. 2002 Jun 15;20(12):2774-82. doi: 10.1200/JCO.2002.07.300. PMID 12065553
- [Background] Wells RJ, Woods WG, Lampkin BC, Nesbit ME, Lee JW, Buckley JD, Versteeg C, Hammond GD. Impact of high-dose cytarabine and asparaginase intensification on childhood acute myeloid leukemia: a report from the Childrens Cancer Group. J Clin Oncol. 1993 Mar;11(3):538-45. doi: 10.1200/JCO.1993.11.3.538. PMID 8445429